CLINICAL TRIAL: NCT00632892
Title: The Correlation Between Oxidative Stress and Indinated Contrast-Media Nephrotoxicity
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: 96013
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-02

CONDITIONS: Kidney Diseases
Keywords: oxidative stress markers in urine; urine norepinephrine; renal tubular enzyme markers
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The urine samples are collected just before and 30 minutes after IVP.The samples are immediately frozen at -80'C until analyzed.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinically, iodinated contrast-medium (CM) is widely used in angiography and computerized tomography. CM-induced nephropathy (CMIN) is one major complication after application of CM. Therefore, how to prevent CMIN is always one of the hot topics concerned by nephrologists, cardiologists, and radiologists.

The present study is aimed to determine the norepinephrine concentration, oxidative markers, and tubular damage markers in the urine samples of patients undergoing intravenous pyelography (IVP).

The working hypothesis is high-osmolarity contrast media (HOCM) causes more oxidative stress and greater tubular damage than iso-osmolarity contrast media (IOCM).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (> 18 years old)
2. Undergoing IVP with an appropriate medical indication
3. Signing informed consent

Exclusion Criteria:

1. Without signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adult patients (> 18 years old)
  2. Undergoing IVP with an appropriate medical indication
  3. Signing informed consent
Sampling Method: Non-Probability Sample
Enrollment: 80
Dates: Start 2007-12; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Pan Chiao, Taipei, Taiwan